CLINICAL TRIAL: NCT01892280
Title: Optimizing Self-Management Adherence and Glycemic Control in Older Teens With Type 1 Diabetes: The Teenwork Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Baylor College of Medicine (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lori Laffel, Chief, Pediatric, Adolescent, & Young Adult Section; Investigator, Genetics & Epidemiology Section, Joslin Diabetes Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2012-11; R01DK095273 (NIH)
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Teenwork Group (Experimental): Teen/family will receive the Teenwork intervention at each quarterly study visit.
  Interventions: Behavioral: Teenwork intervention
- Teenwork/Text Message Group (Experimental): Teen/family will receive the Teenwork intervention at each quarterly study visit. Teen will receive text message reminders to check blood glucose levels at self-selected times.
  Interventions: Behavioral: Teenwork intervention; Behavioral: Text message reminders
- Text Message Group (Experimental): Teen will receive text message reminders to check blood glucose levels at self-selected times.
  Interventions: Behavioral: Text message reminders
- Usual Care Group (No Intervention): Teen/family will receive routine clinical care for the first year of the study (the time period for assessment of primary outcomes). After year 1, teen/family will receive the Teenwork intervention at each remaining study visit and teen will receive text message reminders to check blood glucose levels at self-selected times.

INTERVENTIONS:
Behavioral: Teenwork intervention — Set of psychoeducational modules focused on optimizing diabetes self-care through blood glucose monitoring and insulin administration
  Arms: Teenwork Group; Teenwork/Text Message Group
Behavioral: Text message reminders — Text message reminders to check blood glucose levels at self-selected times
  Arms: Teenwork/Text Message Group; Text Message Group

SUMMARY:
The purpose of this 18-month randomized controlled trial (RCT) is to find out if (1) a set of psychoeducational materials for teens with type 1 diabetes and (2) text message reminders to check blood glucose levels can help improve blood glucose levels in teens with type 1 diabetes.

DETAILED DESCRIPTION:
Glycemic control deteriorates during adolescence as parents become less involved in teens' diabetes management and adherence declines. Thus, there is a need to improve adherence and glycemic control in mid to older teens with type 1 diabetes by strengthening the teens' self-efficacy for daily diabetes self-management to help prepare them for the transition between pediatric and adult care. This 18-month, multi-center RCT is designed to increase frequency of blood glucose monitoring and improve glycemic control in teens with type 1 diabetes through a behavioral intervention called Teenwork with or without text message reminders to check blood glucose levels.

We will implement and evaluate the Teenwork intervention and text message reminders to check blood glucose levels in a 2x2 factorial design in which 300 participants, across two sites, will be randomized to 1 of 4 groups: Teenwork, Text Message, Teenwork/Text Message, or Usual Care.

Participants in the Teenwork Group will meet with a research assistant during each study visit to review strategies for improving self-care, including self-management and self-advocacy, focusing on two areas: blood glucose monitoring and insulin administration. Participants in the Text Message Group will be instructed in the use of the text messaging system. They will receive 2-way text message reminders to check blood glucose levels at self-selected times and to reply by text message with blood glucose results. Participants in the Teenwork/Text Message Group will receive both the Teenwork intervention and the text message reminders (as described above). Participants in the Usual Care Group will receive the same intervention as the Teenwork/Text Message Group, but not until after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Youth age 13-17 years
* Diagnosis of type 1 diabetes according to American Diabetes Association criteria
* Diabetes duration ≥6 months
* Daily insulin dose ≥0.5 units/kg
* A1c ≥6.5%and ≤11%
* Willingness to check blood glucose levels
* Cell phone with text messaging ability
* Clinic attendance

  1. At least one clinic visit at the clinical site in the previous 12 months
  2. Anticipated care at the clinical site for the duration of the study
* Fluency in English (reading, writing, and speaking) for child and parent/guardian
* Enrollment no later than December of the teen's senior year of high school

Exclusion Criteria:

* Pregnancy in the youth participant
* Significant developmental or cognitive disorder that would prevent full study participation
* Significant mental illness, defined by either major psychiatric disorder (e.g., diagnosed eating disorder, major psychoses) or inpatient psychiatric admission within the previous 6 months
* Failure to understand that the 2-way text messaging does NOT result in immediate response from a health care professional; this will be assessed at the time of informed consent/assent
* Participation in another intervention study within the 3 months prior to enrollment
* Other psychosocial, medical, or family issues, as assessed by the teen's pediatric team, that would prevent full study participation

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in glycemic control from baseline to 1 year | Baseline and 1 year
  Glycemic control will be assessed as A1c (DCCT-standardized assay, ref range 4.0-6.0%)

SECONDARY OUTCOMES:
Change in glycemic control from 1 year to 18 months | 1 year and 18 months
  Glycemic control will be assessed as A1c (DCCT-standardized assay, ref range 4.0-6.0%)
Psychosocial factors (self-report surveys) | Baseline, 6 months, 1 year, 18 months
  We will assess psychosocial factors (e.g., diabetes-specific family conflict, diabetes burden, negative affect around blood glucose monitoring, quality of life, depressive symptoms, self-efficacy, disordered eating behaviors) every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori Laffel, MD, MPH, Principal Investigator — Joslin Diabetes Center; Barbara J. Anderson, PhD, Principal Investigator — Texas Children's Hospital/Baylor College of Medicine
Locations (2):
- United States (2):
  - Joslin Diabetes Center, Boston, Massachusetts
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Commissariat PV, Volkening LK, Guo Z, ElBach JL, Butler DA, Laffel LM. Associations between major life events and adherence, glycemic control, and psychosocial characteristics in teens with type 1 diabetes. Pediatr Diabetes. 2018 Feb;19(1):85-91. doi: 10.1111/pedi.12523. Epub 2017 Apr 19. PMID 28425183
- [Result] McGill DE, Volkening LK, Butler DA, Wasserman RM, Anderson BJ, Laffel LM. Text-message responsiveness to blood glucose monitoring reminders is associated with HbA1c benefit in teenagers with Type 1 diabetes. Diabet Med. 2019 May;36(5):600-605. doi: 10.1111/dme.13929. Epub 2019 Feb 25. PMID 30734361
- [Result] Cecilia-Costa R, Volkening LK, Laffel LM. Factors associated with disordered eating behaviours in adolescents with Type 1 diabetes. Diabet Med. 2019 Aug;36(8):1020-1027. doi: 10.1111/dme.13890. Epub 2019 Mar 4. PMID 30582670
- [Result] McGill DE, Laffel LM, Volkening LK, Butler DA, Levy WL, Wasserman RM, Anderson BJ. Text Message Intervention for Teens with Type 1 Diabetes Preserves HbA1c: Results of a Randomized Controlled Trial. Diabetes Technol Ther. 2020 May;22(5):374-382. doi: 10.1089/dia.2019.0350. PMID 32357109
- [Result] Harrington KR, Shapira A, Volkening LK, Butler DA, Anderson BJ, Wasserman RM, Laffel LM. Associations of diabetes self-management characteristics, HbA1c, and psychosocial outcomes with depressive symptoms in a contemporary sample of adolescents with type 1 diabetes. J Diabetes Complications. 2021 Mar;35(3):107838. doi: 10.1016/j.jdiacomp.2020.107838. Epub 2021 Jan 6. PMID 33431226